CLINICAL TRIAL: NCT05244668
Title: Multicenter Validation of the Salivary miRNA Signature of Endometriosis - The ENDOmiARN Salive Test Study
Brief Title: Multicenter Validation of the Salivary miRNA Signature of Endometriosis
Status: Active, not recruiting | Type: Observational
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry); iGenSeq (Unknown)
Responsible Party: Sponsor
Other Study IDs: FR-21-001
Record Dates: First submitted 2022-01-19; First posted 2022-02-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Endometriosis
Keywords: miRNA; MAP; machine learning algorithms
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ENDOmiARN Salive Test is a multicentre external validation study of a salivary signature of endometriosis carried out in France in Obstetrics and Reproductive Medicine departments, in order to evaluate its performance and discuss its use in clinical practice. The clinical application is to significantly reduce the time to diagnosis and improve the care pathway for endometriosis.

The study population is made up of women aged 18 to 43 years with formally diagnosed endometriosis or suspected endometriosis who are already receiving either medical (MAP) or surgical treatment as part of their routine care.

The patients concerned by the study are managed without any change in the care pathway, nor any change in the therapeutic indications, nor any change in the diagnostic examinations (imaging or biology) required according to the context, which are carried out in accordance with the HAS recommendations.

In this study, the management and follow-up of patients :

* Are not imposed by the study: the doctor remains free to make medical prescriptions (treatments and examinations) and to determine the interval between consultation visits,
* Are not modified in comparison with the usual follow-up, except for the performance of :

  * Collection of saliva
  * Electronic collection of the answers to the questionnaires completed by the patient

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 43 years,
* Patient having dated and signed the consent form,
* Patient affiliated to the French health system,
* Patient with pelvic MRI and/or pelvic ultrasound,
* Patient from one of the 3 study populations:

  * Patient with a formal endometriosis diagnosed by clinical examination and imaging AND an indication for specialised endometriosis follow-up or medically assisted procreation (MAP) or surgery validated by RCP (in routine care);
  * Patient with suspected endometriosis for whom the diagnosis is the source of a discrepancy between clinical and radiological data AND a surgical indication validated by RCP (in routine care);
  * Patient with a gynaecological indication for surgery of the small pelvis by laparoscopy or laparoscopy validated in RCP (in routine care) AND symptoms suggestive of endometriosis (dysmenorrhoea, ....)(1).

Exclusion Criteria:

* Patient with recurrence of deep endometriosis (excluding endometrioma),
* Patient with endometriosis of the torus and/or utero-sacral ligaments without indication for surgery,
* Patient with parietal endometriosis alone without indication for surgery,
* Patient with adenomyosis alone on imaging without indication for surgery,
* Patient with gynaecological infection requiring surgical management,
* Pregnant patient,
* Patient infected with the human immunodeficiency virus (HIV),
* Patient with significant difficulties in reading or writing the French language,
* Patient with a personal history of cancer,
* Patient unable to comply with study and/or follow-up procedures,
* Patient who has objected to the collection of her data.
* Patient participating in another clinical research study.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: The study population is made up of women aged 18 to 43 years with a formal diagnosis of endometriosis or suspected endometriosis.
  The patients concerned by the study are already receiving either medical (MAP) or surgical care in a department of Obstetrics and Reproductive Medicine.
  All these patients already benefit from validation of therapeutic indications in a multidisciplinary consultation meeting (medical-surgical or fertility RCP).
  The patients concerned by the study are managed without modification of the care pathway, nor modification of the therapeutic indications, nor modification of the diagnostic examinations (imaging or biology) necessary according to the context, which are carried out according to the recommendations of the HAS.
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
At least a 90% Sensitivity (True Positive Rate) of Endometriosis diagnotic confirmation using a miRNA signature | Through the end of study inclusions, an average of 1 year
  External validation of the salivary signature of endometriosis miRNAs
At least a 90% Specificity (True Negative Rate) of Endometriosis diagnotic confirmation using a miRNA signature | Through the end of study inclusions, an average of 1 year
  External validation of the salivary signature of endometriosis miRNAs

CONTACTS AND LOCATIONS:
Locations (18):
- CHU Québec, Québec, Canada
- France (17):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Alsace
  - CHU de Caen, Caen, Calvados
  - Clinique Tivoli, Bordeaux, Gironde
  - CHU Toulouse - Hôpital Rangueil, Toulouse, Haute Garonne
  - Clinique Pasteur, Toulouse, Haute-Garonne
  - Clinique La Sagesse, Rennes, Ille Et Vilaine
  - Cabinet de Gynécologie Médicale, Lyon, Rhône
  - CHU Rouen, Bois-Guillaume, Seine-Maritime
  - Hôpital BICETRE, Le Kremlin-Bicêtre, Val De Marne
  - Centre médical des Pyramides, Maurepas, Yvelines
  - CHU Angers, Angers
  - CH Bastia, Bastia
  - HCL, Lyon
  - Groupe Hospitalier Saint Josef, Paris
  - Centre d'imagerie Manin Crimée, Paris
  - CHU Tenons, Paris
  - CHU Rennes, Rennes

REFERENCES:
- [Derived] Bendifallah S, Roman H, Suisse S, Spiers A, Petit E, Delbos L, Dabi Y, Touboul C, Dennis T, Merlot B, Sauvanet E, Fauvet R, Jamard E, Clotilde H, Morgane P, Fedida B, Nyangoh K, Lavoue V, Roger CM, Lucas N, Darnaud T, Boudy AS, Genre L, Leguevaque P, Akldios C, Benjoar M, Chantalat E, Tanguy Le Gac Y, Poilblanc M, Rousset P, Fernandez H, Golfier F, Descamps P. Validation of a Saliva Micro-RNA Signature for Endometriosis. NEJM Evid. 2025 Nov;4(11):EVIDoa2400195. doi: 10.1056/EVIDoa2400195. Epub 2025 Oct 28. PMID 41147827
- [Derived] Bendifallah S, Dabi Y, Suisse S, Delbos L, Spiers A, Poilblanc M, Golfier F, Jornea L, Bouteiller D, Fernandez H, Madar A, Petit E, Perotte F, Fauvet R, Benjoar M, Akladios C, Lavoue V, Darnaud T, Merlot B, Roman H, Touboul C, Descamps P. Validation of a Salivary miRNA Signature of Endometriosis - Interim Data. NEJM Evid. 2023 Jul;2(7):EVIDoa2200282. doi: 10.1056/EVIDoa2200282. Epub 2023 Jun 9. PMID 38320163